CLINICAL TRIAL: NCT05464069
Title: A Retrospective Controlled Survey Study to Assess the Safety of Treating Migraine With Nerivio During Pregnancy and 3 Months Postpartum
Brief Title: Safety of Nerivio in Pregnant Women With Migraine
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: TCH011
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2022-06

CONDITIONS: Migraine; Pregnancy Related
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Postpartum females with migraine who used Nerivio during their pregnancy: Postpartum patients with migraine who used Nerivio at least 3 times during their pregnancy. Participants will be recruited from Nerivio's user database
  Interventions: Device: Nerivio
- Postpartum females with migraine who used other migraine therapy during their pregnancy: Postpartum patients with migraine who did not used Nerivio prior and during their pregnancy, and at least 3 months postpartum. Participants will be referred to the study by site co-investigators, who are US-licensed healthcare providers seeing women with headache disorders and/or women during their pre-pregnancy and/or pregnancy period
  Interventions: Drug: Migraine Relief

INTERVENTIONS:
Device: Nerivio — Nerivio is a Remote Electrical Neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application
  Other Names: Neriivo
  Groups: Postpartum females with migraine who used Nerivio during their pregnancy
Drug: Migraine Relief — Any drug for treatment of migraine relief
  Other Names: migraine treatment
  Groups: Postpartum females with migraine who used other migraine therapy during their pregnancy

SUMMARY:
This is a retrospective controlled survey study to assess the safety of treating migraine with Nerivio during pregnancy and 3 months postpartum. The study will compare migraine and pregnancy-related health and baby health between women with migraine who treated migraine attacks during pregnancy with Nerivio (Nerivio group), to women with migraine who did not treat migraine attacks during pregnancy with Nerivio (control group). Nerivio group participants will be recruited from Theranica's user base. Control group participants will be recruited by health care providers, including headache specialists and OBGYNs (study co-investigators). The study is based on an e-Survey including an e-eligibility questionnaire, an e-ICF ande-Questionnaire. Participants will be compensated for their time.

DETAILED DESCRIPTION:
This is a retrospective controlled survey study to assess the safety of treating migraine with Nerivio during pregnancy and 3 months postpartum. The study will compare migraine and pregnancy-related health and baby health between women with migraine who treated migraine attacks during pregnancy with Nerivio (Nerivio group), to women with migraine who did not treat migraine attacks during pregnancy with Nerivio (control group).

Study group: Study group participants will be recruited from Nerivio's user base. An invitation message will be sent via in-app notification and/or email to all Nerivio users who are (1) female, AND (2) between 18 and 42 years of age as of November 1st, 2019 - March 31st, 2021. Users who meet these criteria will be invited to fill in a screening and eligibility questionnaire. If they meet the eligibility criteria, they will be offered the opportunity to participate in the study. Participants will complete and sign an electronic informed consent form. Following consent, participants will be asked to complete the questionnaire. Once complete, participants will be compensated for their time.

Control group: Control group participants will be referred to the study by site co-investigators, who are US-licensed healthcare providers seeing women with headache disorders and/or women during their pre-pregnancy and/or pregnancy period. Patients interested in participating will be directed to the same screening and eligibility questionnaire and will follow the same study design.

Endpoints focus on the health of the mother and the baby, during pregnancy and three months postpartum.

Primary endpoint:

Demonstrate that the study group is not different than the control group in regard to gestational age at delivery (measured in pregnancy weeks).

Secondary endpoints:

Demonstrate that the study group is not different from the control group in:

1. Baby's birth weight (average birth weight)
2. Miscarriage rate (% of miscarriage cases)
3. Preterm birth rate (% cases of preterm pregnancies, as measured in % of pregnancy weeks less than 37)
4. Birth deficits rate (% of birth deficits)
5. Still births rate (% of still births)
6. Meeting developmental milestones following 3 months postnatal (% of babies)
7. Visits to the emergency room or urgent care due to pregnancy and/or migraine symptoms during pregnancy and 3 months postpartum period (# of events)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with migraine
2. History of migraine pre-pregnancy with an average of at least 4 migraine days per month, in the six months prior to the last pregnancy
3. History of pregnancy with last menstrual period (LMP) between November 1st, 2019 - March 31st, 2021. Pregnancy within this time window is the pregnancy of study, termed "study pregnancy"
4. Between 18 and 42 years of age at first day of the last menstrual period (LMP) of "study pregnancy"
5. History of at least 4 migraine attacks during "study pregnancy"
6. In the study group: usage of Nerivio for at least 3 treatments (≥30 minutes/treatment) during "study pregnancy"
7. In the control group: No history of using Nerivio, ever

Exclusion Criteria:

1. History of preterm birth (gestational age at deliver<37 weeks) in previous pregnancies prior to the "study pregnancy"
2. History of congenital malformations or birth defects in previous pregnancies prior to the "study pregnancy"
3. Severe other diseases which started before the "study pregnancy" and lasted into the "study pregnancy" period, including congenital heart disease, arrhythmia, history of myocardial infarction (MI), history of stroke, or active cancer
4. Serious physical injury that occurred during the "study pregnancy": severe car collision injury, serious injury at home/work, etc. Multiple gestation (i.e., pregnancy with more than one baby at a time, such as pregnancy with twins, triplets, and quadruplets) in the "study pregnancy"

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum women
Study Population: Post pregnant women between 18 and 42 years of age at first day of the last menstrual period (LMP) of "study pregnancy."
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, PhD, Principal Investigator — Theranica USA
Locations (2):
- United States (2):
  - University of California San Diego (UCSD), San Diego, California
  - Theranica USA, Montclair, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peretz A, Stark-Inbar A, Harris D, Tamir S, Shmuely S, Ironi A, Halpern A, Chuang L, Riggins N. Safety of remote electrical neuromodulation for acute migraine treatment in pregnant women: A retrospective controlled survey-study. Headache. 2023 Jul-Aug;63(7):968-970. doi: 10.1111/head.14586. Epub 2023 Jun 19. No abstract available. PMID 37335242
- See also: Pubmed reference — https://pubmed.ncbi.nlm.nih.gov/37335242/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Started | 62 | 83
Completed | 59 | 81
Not Completed | 3 | 2
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy | Total
Number analyzed (Participants) | 59 | 81 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (6.1) | 32.2 (6.0) | 32.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 81 | 140
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 46 | 70 | 116
  Black or African American | 2 | 6 | 8
  Asian | 4 | 2 | 6
  Hispanic or Latino | 2 | 1 | 3
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 3 | 1 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — The body Mass Index of the participant prior pregnancy
  Kg/m^2 | 26.8 (7.4) | 25.8 (6.1) | 26.2 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Gestational Age at Delivery
Description: The mean number of gestational age at delivery in both study groups (measured in pregnancy days).
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Measure: Mean (Standard Deviation); unit: Gestational days
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Gestational days | 271 (13) | 273 (9)
Statistical Analysis 1: Comparison: Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy vs Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy; Test type: Superiority; p = 0.160, t-test, 2 sided — Significant level < 0.05

2. Secondary Outcome: Birth Weight
Description: The mean weight of the newborn children at the time of delivery in both study groups (measured in Pounds).
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Measure: Mean (Standard Deviation); unit: Weight (pounds)
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Weight (pounds) | 7.2 (1.2) | 7.2 (1.0)

3. Secondary Outcome: Miscarriage Rate
Description: The percent of miscarriage in both study groups
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Participants | 2 | 3

4. Secondary Outcome: Preterm Birth Rate
Description: The percent of preterm birth (measured in % of pregnancy weeks less than 37) in both study groups
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Participants | 8 | 5

5. Secondary Outcome: Birth Deficits Rate
Description: The percent of birth deficits in both study groups
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Participants | 8 | 11

6. Secondary Outcome: Still Births Rate
Description: The percent of Still birth in both study groups
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Participants | 0 | 0

7. Secondary Outcome: Developmental Milestones Rate Following 3 Months Postnatal
Description: The rate of developmental milestones between the study groups. Develpment milestones includes motor skills, hearing, vision and communication (e.g bringing hands to their mouth, and recognizing familiar voices and faces)
Time Frame: Retrospective Data for up to 55 weeks, collected over 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Participants | 57 | 77

8. Secondary Outcome: Migraine Patterns
Description: The proportion of patients that visits the emergency room or urgent care due to pregnancy and/or migraine symptoms during pregnancy and 3 months postpartum period in both study groups
Time Frame: Retrospective Data for up to 55 weeks, collected over 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
Number analyzed (Participants) | 59 | 81
Participants | 9 | 14

ADVERSE EVENTS:
Time Frame: Retrospective Data for up to 42 weeks, collected over 2 months
Arm/Group | Postpartum Females With Migraine Who Used Nerivio During Their Pregnancy | Postpartum Females With Migraine Who Used Other Migraine Therapy During Their Pregnancy
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/81
Other Adverse Events (participants affected / at risk) | 0/59 | 0/81

LIMITATIONS AND CAVEATS:
1. - The retrospective nature of the study may limit the conclusions of this survey by recall bias
2. - The REN group included 59 patients, making it smaller than groups included in other studies assessing the efficacy and safety of migraine treatments in the general population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT05464069/Prot_SAP_000.pdf